CLINICAL TRIAL: NCT03319784
Title: A Randomized Single Blinded Prospective Analysis for NSAID VS Corticosteroid Shoulder Injection in Diabetic Patients
Brief Title: Analysis for NSAID VS Corticosteroid Shoulder Injection in Diabetic Patients
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: never initiated
Sponsor: Milton S. Hershey Medical Center (Other)
Responsible Party: Principal Investigator, H Mike Kim, Associate Professor of Orthopaedics, Milton S. Hershey Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: STUDY00008014
Record Dates: First submitted 2017-09-16; First posted 2017-10-24 (Actual); Last update posted 2019-02-15 (Actual); Status verified 2019-02

CONDITIONS: Rotator Cuff Tear; Rotator Cuff Injury; Rotator Cuff Tendinitis; Diabetes Mellitus
MeSH Terms: conditions — Rotator Cuff Injuries; Diabetes Mellitus | interventions — Ketorolac; Ketorolac Tromethamine; Triamcinolone Acetonide

STUDY DESIGN:
Who Masked: Participant
Masking Description: Patients will be blinded to the kind of injection they receive, but the physicians who perform the injection will not be blinded for the medical record purposes.
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Ketorolac (Toradol) Injection Group (Active Comparator): Patients will be randomized into two patient groups: Ketorolac (Toradol) injection group (n=30) and or Steroid injection group (n=30). Patients assigned to Ketorolac group will receive a single dose of 60mg of Ketorolac (Toradol) mixed with 8mL of 1% lidocaine with epinephrine 1:100,000. Patients will be blinded to the kind of injection they receive, but the physicians who perform the injection will not be blinded for the medical record purposes. The injection will be done under ultrasound guidance to the subacromial space.
  Interventions: Drug: Ketorolac
- Steroid Injection Group (Active Comparator): Patients will be randomized into two patient groups: Ketorolac (Toradol) injection group (n=30) and or Steroid injection group (n=30). Patients assigned to Steroid group will receive a single dose of 80mg of Triamcinolone Acetonide (Kenalog) mixed with 8mL of 1% lidocaine with epinephrine 1:100,000. Patients will be blinded to the kind of injection they receive, but the physicians who perform the injection will not be blinded for the medical record purposes. The injection will be done under ultrasound guidance to the subacromial space.
  Interventions: Drug: Triamcinolone Acetonide

INTERVENTIONS:
Drug: Ketorolac — Patients assigned to Toradol group will receive a single dose of 60mg of Ketorolac (Toradol) mixed with 8mL of 1% lidocaine with epinephrine 1:100,000.
  Other Names: Toradol
  Arms: Ketorolac (Toradol) Injection Group
Drug: Triamcinolone Acetonide — Patients assigned to Steroid group will receive 80mg of Triamcinolone Acetonide (Kenalog) mixed with 8mL of 1% lidocaine with epinephrine 1:100,000.
  Other Names: Kenalog
  Arms: Steroid Injection Group

SUMMARY:
Sixty patients will be identified in the clinic with rotator cuff tendonitis or a low-grade partial-thickness tear of the rotator cuff that are either insulin-dependent or insulin-independent diabetics. Patients will be informed about the current prospective study and written consent will be obtained. Patient information about kidney function, current diabetic medication type, dose and frequency will be obtained in clinic. If there is a diagnosed kidney function abnormality, the patient will be excluded from the study. Patients will be asked about their most recent HbA1C. If HbA1C has not been checked within the past 3 months, the patient will have HbA1C checked in the lab either same day as the injection or the following day. Patients will be randomized into two patient groups: Toradol (Ketorolac) injection group (n=30) and or Steroid injection group (n=30). The randomization will be done using an online randomization tool: http://www.graphpad.com/quickcalcs/index.cfm.

Patients assigned to Toradol group will receive 60mg of Toradol (Ketorolac) mixed with 8mL of 1% lidocaine with epinephrine 1:100,000. Those assigned to Steroid group will receive 80mg of Kenalog (Triamcinolone Acetonide) mixed with 8mL of 1% lidocaine with epinephrine 1:100,000.

Patients will be blinded to the kind of injection they receive, but the physicians who perform the injection will not be blinded for the medical record purposes. The injection will be done under ultrasound guidance to the subacromial space. Continuous blood glucose measurement will be started in an hour within the injection. An instructional session about continuous glucose monitoring will be given to the patients by our research team immediately following the injection. The blood glucose levels will be monitored for 1 week following the injection. The data will be collected on the patient's return to clinic in 2 weeks. Pain score based on a visual analog scale will be obtained prior to injection, 5 min, 3 days, 1 week, 2 weeks, 4 weeks, 6 weeks, 8 weeks, and 12 weeks after injection. Shoulder range of motion, patient satisfaction, QuickDash score, and ASES survey score will be measured in clinic 4, 8, and 12 weeks after injection.

DETAILED DESCRIPTION:
Day 1: Patient will be seen in the clinic. Patient will be provided information about the study, consented and recruited to the study. Obtain pre-injection HbA1c. If no previous HbA1c, obtain a new one on the following day in the morning Injection will be administered to the patient. Pain score will be obtained prior to injection and 5 min after injection. Blood glucose measurement will be started in an hour of the injection and will last for one week after the injection.

Day 3: Patients will be contacted by phone for pain score.

1 Week: Patients will be contacted by phone for pain score. 2 Weeks: Patient will be seen at clinic for a follow up and for pain score. 4 Weeks: Patient will be seen at clinic for pain score and for range of motion, QuickDASH, and ASES scores.

6 Weeks: Patients will be contacted by phone for pain score. 8 Weeks: Patient will be seen at clinic for pain score and for range of motion, QuickDASH, and ASES scores.

12 Weeks: Patient will be seen at clinic for pain score and for range of motion, QuickDASH, and ASES scores.

ELIGIBILITY:
Inclusion Criteria:

* Patients that are 18 years old or older that have rotator cuff tendinitis and a low-grade partial thickness tear of the rotator cuff confirmed with an imaging study (ultrasound or MRI) with either insulin dependent or insulin independent diabetes.

Exclusion Criteria:

* Patients whom are younger than 18 years old, pregnant women, and prisoners will be excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2018-09-05 (Estimated); Primary Completion 2020-09-05 (Estimated); Study Completion 2020-10-05 (Estimated)

PRIMARY OUTCOMES:
Change in blood glucose level | Participants' blood glucose will be measured 5 minutes after injection and three times daily for one week following injection; Alternatively, using Continuous Glucose Monitoring sensors, blood glucose will be monitored for 1 week following injection.
  The peak and average glucose levels, and duration of the increase will be used as the surrogates of the primary outcome. The peak and average glucose levels will both share the same unit of measure (mg/dL). The duration of the increase will measure the number of hours that the patient experienced an increasing level of glucose.

SECONDARY OUTCOMES:
Visual Analog Scale | Pain scores will be obtained prior to injection, 5 min, 3 days, 1 week, 2 weeks, 4 weeks, 6 weeks, 8 weeks, and 12 weeks after injection.
  Pain scores will be measured using the Visual Analog Scale. Scale: 0 - 10 0 - No pain; 5- Moderate pain; 10 - Extreme pain Lower values = better outcome No subscales will be used
Shoulder Range of Motion | Shoulder range of motion will be measured in clinic 4, 8, and 12 weeks after injection.
Patient Satisfaction | Patient satisfaction will be measured in clinic 4, 8, and 12 weeks after injection.
  Patients will be asked to fill out a questionnaire asking their satisfaction level regarding the treatment.
QuickDASH | QuickDash score will be measured in clinic 4, 8, and 12 weeks after injection.
  The QuickDASH is a shortened version of the DASH (Disabilities of the Arm, Shoulder, and Hand) Outcome Measure. Instead of 30 items, the QuickDASH uses 11 items to measure physical function and symptoms in people with any or multiple musculoskeletal disorders of the upper limb.
American Shoulder and Elbow Surgeon (ASES) Shoulder Score | ASES survey score will be measured in clinic 4, 8, and 12 weeks after injection.
  The ASES questionnaire is composed of both a physician-rated component and a patient-reported component. The patient questions focus on joint pain, instability, and activities of daily living.
  For this study, we will not be using the physician-rated questionnaire and no subscales will be used.
  ASES Patient-rated questionnaire
  Total of 100 maximum points (Weighted 50% for pain and 50% for function) -Higher the score, better the outcome
  Pain portion:
  -The final pain score (maximum 50 points) is calculated by subtracting the Visual Analog Scale (VAS) from 10 and multiplying by five.
  Functional portion:
  * 10 questions rated on a 4-point ordinal scale (from 0-3)
  * Maximum of 30 points. The raw score is multiplied by 5/3 to make the maximal functional score out of 50 possible points. The pain and functional portions are then summed to obtain the final ASES score.

CONTACTS AND LOCATIONS:
Overall Officials: H. Mike Kim, MD, Principal Investigator — Penn State College of Medicine
Locations (1):
- Penn State College of Medicine, Hershey, Pennsylvania, United States